CLINICAL TRIAL: NCT03582215
Title: Assessment of the Human Systemic Absorption of Sunscreen Ingredients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SCR-005
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Systemic Exposure to Sunscreen Ingredients
Keywords: Sunscreen; Pharmacokinetics
MeSH Terms: interventions — avobenzone; octocrylene; terephthalylidene dicamphor sulfonic acid; oxybenzone; homosalate; 2-ethylhexyl salicylate; octylmethoxycinnamate

STUDY DESIGN:
Intervention Model Description: Part 1 of the study has 4 parallel arms where 4 different sunscreen products will be studied. Part 2 of the study has 4 parallel arms where 4 sunscreen products (one from Part 1 and 3 new sunscreen products) will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1: Cream (Experimental): Part 1: Cream
  Ingredients: 2% Avobenzone; 10% Octocrylene; 2% Ecamsule
  Interventions: Drug: Part 1: Cream
- Part 1: Lotion (Experimental): Part 1: Lotion
  Ingredients: 3% Avobenzone; 4% Oxybenzone; 6% Octocrylene
  Interventions: Drug: Part 1: Lotion
- Part 1: Spray 1 (Experimental): Part 1: Spray 1
  Ingredients: 3% Avobenzone; 6% Oxybenzone; 2.35% Octocrylene; 15% Homosalate; 5% Octisalate
  Interventions: Drug: Part 1: Spray 1
- Part 1: Spray 2 (Experimental): Part 1: Spray 2
  Ingredients: 3% Avobenzone; 5% Oxybenzone; 10% Octocrylene
  Interventions: Drug: Part 1: Spray 2
- Part 2: Lotion (Experimental): Part 2: Lotion
  Ingredients: 3% Avobenzone; 4% Oxybenzone; 6% Octocrylene
  Interventions: Drug: Part 2: Lotion
- Part 2: Aerosol Spray (Experimental): Part 2: Aerosol Spray
  Ingredients: 3% Avobenzone; 6% Oxybenzone; 10% Octocrylene; 15% Homosalate; 5% Octisalate
  Interventions: Drug: Part 2: Aerosol Spray
- Part 2: Nonaerosol Spray (Experimental): Part 2: Nonaerosol Spray
  Ingredients: 3% Avobenzone; 10% Octocrylene; 10% Homosalate; 5% Octisalate; 7.5% Octinoxate
  Interventions: Drug: Part 2: Nonaerosol Spray
- Part 2: Pump Spray (Experimental): Part 2: Pump Spray
  Ingredients: 3% Avobenzone; 10% Homosalate; 5% Octisalate; 7.5% Octinoxate
  Interventions: Drug: Part 2: Pump Spray

INTERVENTIONS:
Drug: Part 1: Cream — Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Octocrylene; Ecamsule
  Arms: Part 1: Cream
Drug: Part 1: Lotion — Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Oxybenzone; Octocrylene
  Arms: Part 1: Lotion
Drug: Part 1: Spray 1 — Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Homosalate; Octisalate; Octocrylene; Oxybenzone
  Arms: Part 1: Spray 1
Drug: Part 1: Spray 2 — Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Oxybenzone; Octocrylene
  Arms: Part 1: Spray 2
Drug: Part 2: Lotion — Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Oxybenzone; Octocrylene
  Arms: Part 2: Lotion
Drug: Part 2: Aerosol Spray — Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Oxybenzone; Octocrylene; Homosalate; Octisalate
  Arms: Part 2: Aerosol Spray
Drug: Part 2: Nonaerosol Spray — Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Octocrylene; Homosalate; Octisalate; Octinoxate
  Arms: Part 2: Nonaerosol Spray
Drug: Part 2: Pump Spray — Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
  Other Names: Avobenzone; Homosalate; Octisalate; Octinoxate
  Arms: Part 2: Pump Spray

SUMMARY:
This study is designed to assess the systemic exposure and pharmacokinetics of sunscreen active ingredients (avobenzone, oxybenzone, ecamsule, octocrylene homosalate, octisalate and octinoxate) when sunscreen product is applied under maximal use conditions.

Part 1 is an open-label, randomized, 4-arm study in 24 healthy adult subjects with the primary objective to explore whether the active components (avobenzone, oxybenzone, ecamsule and octocrylene) of 4 sunscreen products (1 sunscreen product in each arm) are absorbed into the systemic circulation when a sunscreen product is applied under maximal use conditions.

One sunscreen product with the highest avobenzone exposure will be selected for the second part of the study. If there is no quantifiable exposure of avobenzone for any of the sunscreen products, the formulation with the highest oxybenzone exposure will be selected for Part 2. In addition, 3 new sunscreen products are included in Part 2.

Part 2 is an open label, 4-arm study in 48 healthy adult subjects with the primary objective to assess the pharmacokinetics of the active components in the selected product from Part 1 and 3 additional products with a combination of active ingredients (avobenzone, oxybenzone, octocrylene, ecamsule homosalate, octisalate and octinoxate as applicable/contained in the different products).

DETAILED DESCRIPTION:
Part 1

Part 1 is an open label, randomized, 4-arm pilot study to evaluate the effects of multiple applications of 4 different topical sunscreen formulations in healthy adult subjects. Each arm will include 6 subjects (3 male and 3 female) with 1 formulation. A total of 24 subjects (12 male and 12 female) from all 4 arms will be admitted to the clinical research unit (CRU) on Day 0. On the morning of Days 1 through 4, subjects will receive a topical application of the study drug at approximately 0900 hours. The study product will be weighed in advance and applied by a qualified person from the study team. Subjects will then receive 3 more topical applications on the same day at 2, 4, and 6 hours after the first dose.

Part 2

Part 2 is an open label, 4-arm study to evaluate the pharmacokinetics of avobenzone, oxybenzone, octocrylene, ecamsule homosalate, octisalate and octinoxate (as applicable in the different products) after multiple applications of a topical sunscreen formulation in healthy adult subjects. Part 2 will include 48 subjects (24 male and 24 female) and each arm will include 12 subjects (6 male and 6 female). One of the formulations in Part 2 will be selected based on the plasma exposure data from the pilot study (Part 1). A total of 48 subjects (24 male and 24 female) will be admitted to the CRU on Day 0. On the morning of Days 1 through 4, subjects will receive a topical application of the study product at approximately 0900 hours. The study drug will be weighed in advance and applied by a qualified person from the study team. Subjects will only receive one application on Day 1. On Days 2, 3 and 4 subjects will receive an initial dose and 3 more topical applications on the same day at 2, 4, and 6 hours after the first dose.

Parts 1 and 2

In both parts, approximately 2 mg of active sunscreen ingredient per 1 cm2 of body surface (calculation per method of Dubois) will be evenly applied 4 times per study day (except for a one-time application on the first day in part 2) to areas of the body typically exposed to the sun: face, ears, neck, torso, arms, and legs (approximately 75% of the body surface area). The antecubital areas will be avoided when applying the sunscreen due to potential contamination of the sites used for intravenous pharmacokinetic (PK) blood sample collection. The topical applications of study drug will be administered with subjects in swim wear to simulate real world settings as well as for easy application. In addition to swim wear, subjects may wear scrubs in between applications and at other times throughout the day/night. Subjects are required to shower each morning after the first PK blood sample collection (and before the first dose of the day), but not at other times during the day.

Blood samples (approximately 10 mL per sample) will be collected for determination of plasma concentrations for all active ingredients (avobenzone, oxybenzone, octocrylene, ecamsule, homosalate, octisalate and octinoxate, where applicable).

Safety evaluations will include adverse event (AE) monitoring, vital sign measurements, and physical examinations. All AEs reported by the subject or observed by the investigator or clinical research unit (CRU) staff will be recorded. Any AE reported after the informed consent is signed and before study drug application will be recorded as medical history.

Subjects will remain in the CRU after admission on Day 0 until the morning of Day 7 following completion of scheduled end-of-study activities for Part 1. For Part 2, subjects will undergo the same schedule but will return to the clinic for follow-up visits on Days 10, 14 and 21. Subjects will then be discharged following completion of End-of-Study activities.

Subjects are not allowed to use products containing any of these active ingredients from 7 days before check-in until completion of End-of-Study procedures.

ELIGIBILITY:
Subjects who meet all of the following inclusion criteria will be eligible to participate in the study:

1. Subject signs an institutional review board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 60 years of age, inclusive, who has a body mass index of 18.5 to 29.9 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and Check-in (Day 0).
5. Subject has no known or suspected allergies or sensitivities to any components of the sunscreen formulation.
6. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before Check in (Day 0) and agree to remain strictly abstinent for the duration of the study and for at least 1 month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day 0) until at least 1 month after the last application of study drug.
7. Female subjects must not be pregnant or lactating before enrollment in the study.
8. Male subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day 0) until at least 1 month after the last application of study drug.
9. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Note: subjects with any skin type or skin pigment type may be eligible for the study.

Subjects who meet any of the following exclusion criteria will not be eligible to participate in the study:

1. Subject has broken, irritated, or unhealed skin.
2. Subject has an active sunburn.
3. Subject has used a tanning bed in the previous 4 weeks.
4. Subject has known skin or autoimmune disease(s).
5. Subject is anemic or has any chronic condition(s) that may impact blood sample collection.
6. Subject has any underlying disease or surgical or medical condition (e.g., cancer, human immunodeficiency virus [HIV], severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study.
7. Subject has known or suspected allergies or sensitivities to any components of the sunscreen formulation.
8. Subject has clinical laboratory test results (hematology and serum chemistry) at Screening that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
9. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
10. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
11. Subject has received or applied the topical sunscreen formulations used in the current study, or any other product containing the active ingredients of the topical sunscreen formulations used in the current study, within 7 days before Check in (Day 0).
12. Subject has used any personal care product(s) containing any active sunscreen ingredient, such sunscreen products, hand or body moisturizing lotion, makeup or foundation, lip balm, or lipstick, within 7 days before Check in (Day 0).
13. Subject is unable or unwilling to tolerate the scent of sunscreen for the duration of the treatment period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the clinical study was included as part of supplementary materials for both publications
Supporting Information: Study Protocol, CSR
Time Frame: Jan 2020 - supplementary materials included with publications
Access Criteria: Access to JAMA. De-identified data has been included under supplement 3 for Part 1 (Matta et al, 2019 JAMA) and Part 2 (Matta et al, 2020, JAMA) of this clinical study
  Part 1 study data:
  https://cdn.jamanetwork.com/ama/content_public/journal/jama/938034/jpc190002supp3_prod.xlsx

REFERENCES:
- [Result] Matta MK, Zusterzeel R, Pilli NR, Patel V, Volpe DA, Florian J, Oh L, Bashaw E, Zineh I, Sanabria C, Kemp S, Godfrey A, Adah S, Coelho S, Wang J, Furlong LA, Ganley C, Michele T, Strauss DG. Effect of Sunscreen Application Under Maximal Use Conditions on Plasma Concentration of Sunscreen Active Ingredients: A Randomized Clinical Trial. JAMA. 2019 Jun 4;321(21):2082-2091. doi: 10.1001/jama.2019.5586. PMID 31058986
- [Result] Matta MK, Florian J, Zusterzeel R, Pilli NR, Patel V, Volpe DA, Yang Y, Oh L, Bashaw E, Zineh I, Sanabria C, Kemp S, Godfrey A, Adah S, Coelho S, Wang J, Furlong LA, Ganley C, Michele T, Strauss DG. Effect of Sunscreen Application on Plasma Concentration of Sunscreen Active Ingredients: A Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):256-267. doi: 10.1001/jama.2019.20747. PMID 31961417
- [Derived] Najjar A, Schepky A, Krueger CT, Dent M, Cable S, Li H, Gregoire S, Roussel L, Noel-Voisin A, Hewitt NJ, Cardamone E. Use of Physiologically-Based Kinetics Modelling to Reliably Predict Internal Concentrations of the UV Filter, Homosalate, After Repeated Oral and Topical Application. Front Pharmacol. 2022 Jan 4;12:802514. doi: 10.3389/fphar.2021.802514. eCollection 2021. PMID 35058784

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Equal allocation of men and women for each treatment arm.
Groups:
- Part 1: Cream: Part 1: Cream:
  Ingredients: 2% Avobenzone; 10% Octocrylene; 2% Ecamsule
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 1: Lotion: Part 1: Lotion:
  Ingredients: 3% Avobenzone; 4% Oxybenzone; 6% Octocrylene
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 1: Spray 1: Part 1: Spray 1:
  Ingredients: 3% Avobenzone; 6% Oxybenzone; 2.35% Octocrylene; 15% Homosalate; 5% Octisalate
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 1: Spray 2: Part 1: Spray 2:
  Ingredients: 3% Avobenzone; 5% Oxybenzone; 10% Octocrylene
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 2: Lotion: Part 2: Lotion:
  Ingredients: 3% Avobenzone; 4% Oxybenzone; 6% Octocrylene
  One sunscreen product with the highest avobenzone exposure will be selected for the second part of the study. If there is no quantifiable exposure of avobenzone for any of the sunscreen products, the formulation with the highest oxybenzone exposure will be selected for Part 2.
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
- Part 2: Aerosol Spray: Part 2: Aerosol Spray:
  Ingredients: 3% Avobenzone; 6% Oxybenzone; 10% Octocrylene; 15% Homosalate; 5% Octisalate
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
- Part 2: Nonaerosol Spray: Part 2: Nonaerosol Spray:
  Ingredients: 3% Avobenzone; 10% Octocrylene; 10% Homosalate; 5% Octisalate; 7.5% Octinoxate
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
- Part 2: Pump Spray: Part 2: Pump Spray:
  Ingredients: 3% Avobenzone; 10% Homosalate; 5% Octisalate; 7.5% Octinoxate
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
Period: Overall Study
Arm/Group | Part 1: Cream | Part 1: Lotion | Part 1: Spray 1 | Part 1: Spray 2 | Part 2: Lotion | Part 2: Aerosol Spray | Part 2: Nonaerosol Spray | Part 2: Pump Spray
Started | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12
Completed | 5 | 6 | 6 | 6 | 12 | 12 | 10 | 10
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Cream: Part 1: Cream
  Ingredients: 2% Avobenzone; 10% Octocrylene; 2% Ecamsule
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 1: Lotion: Part 1: Lotion
  Ingredients: 3% Avobenzone; 4% Oxybenzone; 6% Octocrylene
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 1: Spray 1: Part 1: Spray 1
  Ingredients: 3% Avobenzone; 6% Oxybenzone; 2.35% Octocrylene; 15% Homosalate; 5% Octisalate
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 1: Spray 2: Part 1: Spray 2
  Ingredients: 3% Avobenzone; 5% Oxybenzone; 10% Octocrylene
  Approximately 2 mg per cm2 of body surface will be applied topically 4 times per day for 4 days to approximately 75% of the body surface area
- Part 2: Lotion: Part 2: Lotion
  Ingredients: 3% Avobenzone; 4% Oxybenzone; 6% Octocrylene
  One sunscreen product with the highest avobenzone exposure will be selected for the second part of the study. If there is no quantifiable exposure of avobenzone for any of the sunscreen products, the formulation with the highest oxybenzone exposure will be selected for Part 2.
  Part 2: Sunscreen Product #1, 2, 3 or 4: Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
- Part 2: Aerosol Spray: Part 2: Aerosol Spray
  Ingredients: 3% Avobenzone; 6% Oxybenzone; 10% Octocrylene; 15% Homosalate; 5% Octisalate
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
- Part 2: Nonaerosol Spray: Part 2: Nonaerosol Spray
  Ingredients: 3% Avobenzone; 10% Octocrylene; 10% Homosalate; 5% Octisalate; 7.5% Octinoxate
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
- Part 2: Pump Spray: Part 2: Pump Spray
  Ingredients: 3% Avobenzone; 10% Homosalate; 5% Octisalate; 7.5% Octinoxate
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
- Total: Total of all reporting groups
Arm/Group | Part 1: Cream | Part 1: Lotion | Part 1: Spray 1 | Part 1: Spray 2 | Part 2: Lotion | Part 2: Aerosol Spray | Part 2: Nonaerosol Spray | Part 2: Pump Spray | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (10.8) | 34.5 (6.9) | 42.8 (13.0) | 33.7 (9.1) | 45.1 (13.8) | 41.4 (13.4) | 39.2 (12.2) | 29.0 (8.5) | 37.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 36
  Male | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 7
  Not Hispanic or Latino | 5 | 5 | 4 | 6 | 11 | 11 | 12 | 11 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 1 | 4 | 4 | 5 | 4 | 10 | 37
  White | 0 | 2 | 5 | 2 | 8 | 7 | 6 | 2 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12 | 72
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 26.7 (2.8) | 25.4 (2.5) | 24.1 (3.2) | 24.0 (3.0) | 26.2 (2.2) | 25.8 (3.7) | 25.8 (2.4) | 26.0 (3.3) | 25.7 (2.9)
Fitzpatrick Skin Type [Number; unit: participants] — Type I - highly sensitive, always burns, never tans (e.g. Red hair with freckles); Type II - Very sun sensitive, burns easily, tans minimally (e.g. Fair skinned, fair haired Caucasians); Type III - Sun sensitive skin, sometimes burns, slows tans to light brown (e.g. Darker Caucasians); Type IV - Minimally sun sensitive, burns minimally, always tans to moderate brown (e.g. Mediterranean type Caucasians, some Hispanics); Type V - Sun insensitive skin, rarely burns, tans well (e.g. Some Hispanics, some Blacks); and Type VI - Sun insensitive, never burns, deeply pigmented (e.g. Darker Blacks).
  participants
    I | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    II | 0 | 0 | 1 | 0 | 3 | 2 | 3 | 1 | 10
    III | 0 | 1 | 3 | 1 | 5 | 10 | 6 | 9 | 35
    IV | 0 | 3 | 0 | 1 | 4 | 0 | 3 | 2 | 13
    V | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 8
    VI | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 6
Weight (kg) [Mean (Standard Deviation); unit: kg] | 77.6 (10.4) | 73.2 (17.3) | 70.9 (9.9) | 69.1 (12.5) | 76.3 (10.8) | 76.0 (15.6) | 72.0 (8.9) | 75.5 (12.9) | 74.2 (12.1)
Height (cm) [Mean (Standard Deviation); unit: cm] | 170.7 (9.9) | 168.4 (15.5) | 70.9 (9.9) | 171.7 (6.0) | 170.3 (9.7) | 171.0 (11.0) | 167.0 (9.3) | 170.2 (11.1) | 169.8 (10.0)
Body surface area (m^2) [Mean (Standard Deviation); unit: m^2] | 1.9 (0.2) | 1.8 (0.3) | 1.8 (0.1) | 1.8 (0.2) | 1.9 (0.2) | 1.9 (0.2) | 1.8 (0.2) | 1.9 (0.2) | 1.9 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Avobenzone Maximum Concentration
Description: Maximum concentration (observed peak drug concentration) (Cmax)
Time Frame: 0, 0.5, 1, 1.5, 2, 4, 6, 8, 9, 10, 12, 14, 23, 28, 33, 47, 52, 57, 71, 73, 74, 76, 78, 81, 82, 84, 86, 95, 120, and 144 h for Part 1; same time points and 216, 312, and 480 h for Part 2
Population: All subjects who received at least one application and had at least one pharmacokinetic sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cream | Part 1: Lotion | Part 1: Spray 1 | Part 1: Spray 2 | Part 2: Lotion | Part 2: Aerosol Spray | Part 2: Nonaerosol Spray | Part 2: Pump Spray
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12
ng/mL | 1.8 (32) | 4.3 (46) | 4.0 (61) | 3.4 (77) | 7.1 (74) | 3.5 (71) | 3.5 (73) | 3.3 (48)

2. Secondary Outcome: Oxybenzone Maximum Concentration
Description: Maximum concentration (observed peak drug concentration) (Cmax)
Time Frame: as for outcome 1
Population: All subjects who received at least one application and had at least one pharmacokinetic sample. For Part 1, cream and for Part 2, nonaerosol spray and pump spray products did not contain oxybenzone and were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Lotion | Part 1: Spray 1 | Part 1: Spray 2 | Part 2: Lotion | Part 2: Aerosol Spray
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 12
ng/mL | 169.3 (45) | 209.6 (67) | 194.9 (52) | 258.1 (53) | 180.1 (57)

3. Secondary Outcome: Octocrylene Maximum Concentration
Description: Maximum concentration (observed peak drug concentration) (Cmax)
Time Frame: as for outcome 1
Population: All subjects who received at least one application and had at least one pharmacokinetic sample. For Part 2, pump spray product did not contain octocrylene and was excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cream | Part 1: Lotion | Part 1: Spray 1 | Part 1: Spray 2 | Part 2: Lotion | Part 2: Aerosol Spray | Part 2: Nonaerosol Spray
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 12 | 12
ng/mL | 5.7 (47) | 5.7 (66) | 2.9 (102) | 7.8 (113) | 7.8 (87) | 6.6 (78) | 6.6 (104)

4. Secondary Outcome: Ecamsule Maximum Concentration
Description: Maximum concentration (observed peak drug concentration) (Cmax)
Time Frame: 0, 0.5, 1, 1.5, 2, 4, 6, 8, 9, 10, 12, 14, 23, 28, 33, 47, 52, 57, 71, 73, 74, 76, 78, 81, 82, 84, 86, 95, 120, and 144 h for Part 1
Population: All subjects who received at least one application and had at least one pharmacokinetic sample. For Part 1, lotion, spray 1, and spray 2 and for Part 2, lotion, aerosol spray, nonaerosol spray, and pump spray did not contain ecamsule and were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cream
Number analyzed (Participants) | 6
ng/mL | 1.5 (166)

5. Secondary Outcome: Homosalate Maximum Concentration
Description: Maximum concentration (observed peak drug concentration) (Cmax)
Time Frame: 0, 0.5, 1, 1.5, 2, 4, 6, 8, 9, 10, 12, 14, 23, 28, 33, 47, 52, 57, 71, 73, 74, 76, 78, 81, 82, 84, 86, 95, 120, 144, 216, 312, and 480 h for Part 2
Population: All subjects who received at least one application and had at least one pharmacokinetic sample. For Part 1, cream, lotion, and spray 2 and for Part 2, lotion did not contain homosalate and were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Spray 1 | Part 2: Aerosol Spray | Part 2: Nonaerosol Spray | Part 2: Pump Spray
Number analyzed (Participants) | 6 | 12 | 12 | 12
ng/mL | 40.3 (74) | 23.1 (68) | 17.9 (62) | 13.9 (70)

6. Secondary Outcome: Octisalate Maximum Concentration
Description: Maximum concentration (observed peak drug concentration) (Cmax)
Time Frame: as for outcome 5
Population: All subjects who received at least one application and had at least one pharmacokinetic sample. For Part 1, cream, lotion, and spray 2 and for Part 2, lotion did not contain octisalate and were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Spray 1 | Part 2: Aerosol Spray | Part 2: Nonaerosol Spray | Part 2: Pump Spray
Number analyzed (Participants) | 6 | 12 | 12 | 12
ng/mL | 10.0 (46) | 5.1 (82) | 5.8 (77) | 4.6 (98)

7. Secondary Outcome: Octinoxate Maximum Concentration
Description: Maximum concentration (observed peak drug concentration) (Cmax)
Time Frame: as for outcome 5
Population: All subjects who received at least one application and had at least one pharmacokinetic sample. For Part 1, octinoxate was not analyzed for cream, lotion, spray 1, and spray 2 and all products were excluded from the analysis. For Part 2, lotion and aerosol spray did not contain octinoxate and were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Nonaerosol Spray | Part 2: Pump Spray
Number analyzed (Participants) | 12 | 12
ng/mL | 7.9 (87) | 5.2 (68)

ADVERSE EVENTS:
Time Frame: 7 days for part 1; 21 days for part 2
Description: MedDRA
Groups:
- Part 2: Lotion: Part 2: Lotion
  Ingredients: 3% Avobenzone; 4% Oxybenzone; 6% Octocrylene
  Approximately 2 mg per cm2 of body surface will be applied topically 1 time on day 1 and 4 times per day on following 3 days to approximately 75% of the body surface area
Arm/Group | Part 1: Cream | Part 1: Lotion | Part 1: Spray 1 | Part 1: Spray 2 | Part 2: Lotion | Part 2: Aerosol Spray | Part 2: Nonaerosol Spray | Part 2: Pump Spray
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/6 | 3/6 | 1/6 | 2/6 | 6/12 | 9/12 | 11/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cream (N=6) | Part 1: Lotion (N=6) | Part 1: Spray 1 (N=6) | Part 1: Spray 2 (N=6) | Part 2: Lotion (N=12) | Part 2: Aerosol Spray (N=12) | Part 2: Nonaerosol Spray (N=12) | Part 2: Pump Spray (N=12)
Abodinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye burning (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 6 (7) | 5 (11) | 2 (7)
Application site erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 0 (0)
Burning sensation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel punctue site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was conducted in indoor conditions and was not designed to assess differences by formulation or participant factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT03582215/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03582215/SAP_001.pdf